CLINICAL TRIAL: NCT00565539
Title: A Phase 1 Study to Assess the Safety and Antiviral Activity of PEG-rIL-29 Administered as a Single Agent and in Combination With Ribavirin in Treatment-Relapsed and Treatment-Naive Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Study of PEG-rIL-29 (or PEG-IFN Lambda) in Subjects With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Sherri Souza, Clinical Trial Manager, ZymoGenetics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 526F06
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Hepatitis C, Chronic
Keywords: PEGylated recombinant interleukin 29; interferon lambda; interleukin 29; hepatitis C; virus; infection; liver
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Virus Diseases; Infections | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PEGylated recombinant interleukin 29 (PEG-rIL-29) — subcutaneous administration either weekly or every other week
  Other Names: PEGylated interferon lambda (PEG-IFN lambda)

SUMMARY:
Interleukin 29 (IL-29) is a substance that is produced in the body to help fight viral infections. The purpose of this study is to test the safety and antiviral effects of PEG-rIL-29 (a man-made form of IL-29) when it is given either by itself at different doses or in combination with the approved dose of ribavirin (an antiviral drug) to subjects with hepatitis C infection who have received no prior treatment for this disease or who have relapsed following previous treatment with PEGylated interferon alpha (PEG-IFN-α), or other form of IFN-α, and ribavirin.

DETAILED DESCRIPTION:
This is a 3-part study of PEG-rIL-29 in subjects with chronic genotype 1 hepatitis C virus infection who have either received no prior treatment with a PEGylated IFN-α (or other form of IFN-α) or who have relapsed following prior treatment with a PEGylated IFN-α (or other form of IFN-α) and ribavirin. Part 1 of the study will evaluate the safety and tolerability of escalating doses of PEG-rIL-29 when given as a single agent either every other week or weekly over a 4-week period to treatment-relapsed subjects. Part 2 of the study will evaluate dose levels and/or schedules of PEG-rIL-29 in combination with daily oral ribavirin administered over a 4-week period to treatment-relapsed subjects. Part 3 of the study will evaluate dose levels and/or schedules of PEG-rIL-29 in combination with daily oral ribavirin administered over a 4-week period to subjects who have received no prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed subjects (Parts 1 and 2) -- Prior treatment for HCV with PEG-IFN-alpha (or other IFN-alpha) and ribavirin for at least 12 weeks. Naive subjects (Part 3) -- No prior treatment with PEG-IFN-alpha (or other IFN-alpha)
* Genotype 1 HCV RNA greater than or equal to 100,000 IU/mL. Mixed genotype HCV infection is not allowed
* Documented liver biopsy ≤2 years of study enrollment with Ishak score ≤4
* No evidence of hepatocellular carcinoma documented by abdominal imaging within 12 months of study entry
* no evidence of clinically significant diastolic or systolic dysfunction or other clinically significant abnormalities on echocardiogram or ECG
* Negative drug and alcohol tests except for physician prescribed or approved medication
* If male, or female of child-bearing potential, agrees to use 2 forms of medically accepted contraception while on study

Exclusion Criteria:

* Evidence of decompensated liver disease
* History of hypersensitivity to IFN-alpha or ribavirin
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous 6 months
* Undergone surgery or received blood products within 30 days prior to study enrollment
* Prior history of cardiomyopathy, coronary artery disease including angina, interventive procedure for coronary artery disease including angioplasty, stent procedure or cardiac bypass surgery, prior myocardial infarction, or ventricular tachycardia
* Prior or current history of hemoglobinopathy or hemolytic anemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Adverse events and standard clinical laboratory abnormalities | Day 59

SECONDARY OUTCOMES:
HCV RNA levels, serum concentrations of PEG-rIL-29, serum beta2-microglobulin (B2M) levels, serum 2'5' oligoadenylate synthetase (OAS) levels, the presence of anti-PEG-rIL-29 antibodies | Day 59

CONTACTS AND LOCATIONS:
Overall Officials: Diana F Hausman, MD, Study Director — ZymoGenetics
Locations (11):
- United States (10):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University Hospital (UMDNJ), Newark, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - Michael E. DeBakey Veterans Affairs Medical Center, Baylor College of Medicine, Houston, Texas
  - St. Luke's Advanced Liver Therapies, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - VCUHS Hepatology Research Division, Richmond, Virginia
- London Health Sciences Center, London, Ontario, Canada